CLINICAL TRIAL: NCT01689649
Title: Open Flexible Dose Optimisation Trial Assessing Tolerability and Efficacy of Topiramate Monotherapy in Recently Diagnosed Patients With Epilepsy Who Are Treatment Naive or Have Failed One Anti-Epileptic Drug Treatment in Monotherapy
Brief Title: A Study to Assess Tolerability and Efficacy of Topiramate Monotherapy in Recently Diagnosed Patients With Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017830; TOPMATEPY4049 (Other: Janssen-Cilag VIETNAM); TOP-VN -0107 (Other: Janssen-Cilag VIETNAM)
Record Dates: First submitted 2012-08-23; First posted 2012-09-21 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizures; Topiramate; Anti-epileptic drug; Nervous disorder
MeSH Terms: conditions — Epilepsy; Seizures; Nervous System Diseases | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Topiramate (Experimental): For children: Children will start on topiramate with a dosage of 0.5mg/kg in the evening, followed by 0.5mg/kg/day weekly increments until an initial target dose of 3mg/kg/day is reached. The total daily topiramate dose for children may, not exceed 9mg/kg/day. For adult patients: Adult patients start on topiramate with a dosage of 25mg/day in the evening, followed by weekly increments of 25 mg/day until an initial target dose of 100mg/day is reached. The dose of topiramate may be increased to the optimal dose with weekly increments of 0.5mg/kg/day and of 25 mg/day for children and adults, respectively at the discretion of the investigator.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — The patients will receive topiramate tablet twice daily orally up to 16 weeks.

SUMMARY:
The purpose of this dose optimization study is to assess tolerability and efficacy of topiramate monotherapy in recently diagnosed patients with epilepsy who are treatment naive or have failed one anti-epileptic drug (AED) treatment in monotherapy.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), dose optimization trial to assess the tolerability and efficacy of topiramate as monotherapy in recently (within 5 years) diagnosed patients with epilepsy. Treatment naive patients (patients who have never received the treatment before) and patients who failed on their first AED in monotherapy are allowed. Failure is defined as a lack of efficacy and/or tolerability of that AED and the reason for failure is recorded by the physician. A lack of efficacy is characterized when the patient has been treated with AED at target dose but the patient still has seizure. Topiramate will first be titrated up to an initial target dose that will be reached after 4-6 weeks. Further dose titration is guided by the clinical response of the individual patient, but the dose may not exceed a maximum of 400mg/day [9mg/kg/day for children]. If the patient uses an AED at entry, the AED will be fully tapered off over a period of 3 weeks, starting at the beginning of week 2, in order to have all patients on topiramate monotherapy at visit 3. Tapering the AED off may, however, extend this 3-week period if clinically indicated. Visits will be performed at baseline and after 2, 4, 8, 12, 16 weeks. The total duration for each patient in the study will be 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Has been diagnosed with epilepsy within the past 5 years with Primary Generalized Tonic-Clonic (PGTC) seizures as well as partial onset seizures with or without secondary generalization
* Therapy naive, or being treated with their first anti-epileptic drug (AED) in monotherapy that fails in efficacy, tolerability, or both, and not in need of a combination AED therapy
* Informed Assent in children at least 7 years and older

Exclusion Criteria:

* Have pseudoseizures or the treatable cause of the seizures (eg, metabolic disorder, toxic exposure, active infection or neoplasia)
* Has any clinically relevant progressive or serious illness (eg, liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, psychiatric, or metabolic disturbance)
* Pregnant or breast-feeding
* Has a history or suspicion of alcohol or drug abuse
* Must have on current treatment with furosemide, hydrochlorothiazide, monoamine oxidase inhibitors

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 139 (Actual)
Dates: Start 2008-05-02 (Actual); Primary Completion 2010-01-19 (Actual); Study Completion 2010-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag VIETNAM Clinical Trial, Study Director — Janssen-Cilag VIETNAM
Locations (2):
- Vietnam (2):
  - Hanoi
  - Hochiminh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 139 epileptic participants from three participating centers (Neurological department of the Central (Vietnam-Sweden) Pediatrics Hospital, Neurological department of Children's Hospital N0 II at Ho Chi Minh City and the Children's Outpatient Clinic of the Mental Hospital at Ho Chi Minh City) were enrolled in this study to receive topiramate.
Pre-assignment Details: Out of 139 participants, 132 participants were included in the safety analysis, 117 participants completed the trial, entering efficacy analysis and 22 participants were withdrawn from the study.
Groups:
- Topiramate: The participants will receive an initial dose of 0.5mg/kg per oral in the evening, followed by increasing dosage of 0.5 mg/kg/day every week during 6 weeks until the target dose of 3 mg/kg/day being achieved. Subsequent dose is titrated by increasing 0.5 mg/kg/day every week to reach optimal dose according to efficacy and tolerability, but not exceeding total dose of 9 mg/kg/day.
Period: Overall Study
Arm/Group | Topiramate
Started | 139
Completed | 117
Not Completed | 22
Not completed — Lack of Efficacy | 3
Not completed — Non-compliance | 11
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Topiramate
Number analyzed (Participants) | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (3.1) [4 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Wiith Reduction in Number of Seizures Greater Than or Equal to 50%, During the Last 4 Months of Treatment
Time Frame: Month 1, Month 3 and Month 4
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 139
percentage of participants
  Month 1 | 7.0
  Month 3 | 2.4
  Month 4 | 3.0

2. Primary Outcome: Percentage of Participants Wiith Reduction in Number of Seizures Greater Than or Equal to 75%, During the Last 4 Months of Treatment
Time Frame: Month 1, Month 3 and Month 4
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 139
percentage of participants
  Month 1 | 20.3
  Month 3 | 16.9
  Month 4 | 16.0

3. Primary Outcome: Percentage of Seizure Free Participants During the Last 4 Months of Treatment
Time Frame: Month 1, Month 3 and Month 4
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 139
percentage of participants
  Month 1 | 58.6
  Month 3 | 67.0
  Month 4 | 70.0

4. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 50%, 75% and 100% Reduction in Seizures as Per the Seizure Types (Partial, Secondarily Generalized and Generalized Tonic and Clonic Siezures) After 16 Weeks
Time Frame: Month 1, Month 3 and Month 4
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 139
percentage of participants
  Partial seizures with ≥50% | 3.0
  Secondarily generalized seizure with ≥50% | 3.3
  Generalized tonic clonic seizure with ≥50% | 2.0
  Partial seizures with ≥75% | 17.5
  Secondarily generalized seizure with ≥75% | 26.7
  Generalized tonic clonic seizure with ≥75% | 10.0
  Partial seizures with 100% | 65.0
  Secondarily generalized seizure with 100% | 60.0
  Generalized tonic clonic seizure with 100% | 80.0

5. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 50%, 75% and 100% Reduction in Seizures as Per the Seizure Frequency (Less Than 4, 4 to 10 and Greater Than 10) After 16 Weeks
Time Frame: Month 4
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 139
percentage of participants
  < 4 seizures/month with ≥50% | 3.0
  < 4 seizures/month with ≥75% | 5.7
  < 4 seizures/month 100% | 74.3
  4-10 seizures/month with ≥50% | 5.7
  4-10 seizures/month with ≥75% | 11.0
  4-10 seizures/month with 100% | 71.0
  >10 seizures/month with ≥50% | 0.0
  >10 seizures/month with ≥75% | 28.0
  >10 seizures/month with 100% | 66.0

6. Secondary Outcome: General Clinical Assessment Before and After Treatment
Description: The general clinical assessment is measured by clinical global impression scale. The scale is used to grade the participants as very good, good, fairly good, medium and Poor before (Visit 1) and after treatment (Visit 6).
Time Frame: Baseline (Day 0) and Month 4
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 139
percentage of participants
  Visit 1: Very good | 0.0
  Visit 6: Very good | 17.9
  Visit 1: Good | 1.4
  Visit 6: Good | 52.8
  Visit 1: Fairly good | 37.7
  Visit 6: Fairly good | 25.2
  Visit 1: Medium | 44.9
  Visit 6: Medium | 1.6
  Visit 1: Poor | 15.9
  Visit 6: Poor | 2.4

7. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 50%, 75% and 100% Reduction in Seizures With or Without Previous Treatment
Time Frame: Month 4
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 139
percentage of participants
  WIth previous treatment ≥50% | 2.3
  WIth previous treatment ≥75% | 11.4
  WIth previous treatment 100% | 70.5
  WIthout previous treatment ≥50% | 2.7
  WIthout previous treatment ≥75% | 19.2
  WIthout previous treatment 100% | 69.9

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Out of 139 participants, 132 participants were included in the safety analysis, 117 participants completed the trial, entering efficacy analysis and 22 participants were withdrawn from the study.
Groups:
- Topiramate: The participants will receive an initial dose of 0.5mg/kg per oral (PO) in the evening, followed by increasing dosage of 0.5 mg/kg/day every week during 6 weeks until the target dose of 3 mg/kg/day being achieved. Subsequent dose is titrated by increasing 0.5 mg/kg/day every week to reach optimal dose according to efficacy and tolerability, but not exceeding total dose of 9 mg/kg/day.
Arm/Group | Topiramate
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 57/132
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=132)
Fever (General disorders) | 10
Weight loss (General disorders) | 30
Anorexia (General disorders) | 16
Mood disorder (Psychiatric disorders) | 3
Attention disorder (Psychiatric disorders) | 3
Infection (Infections and infestations) | 8
Sleep disorder (Psychiatric disorders) | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 8
Headache (Nervous system disorders) | 5
Itching (Skin and subcutaneous tissue disorders) | 4
Urinary frequency (Renal and urinary disorders) | 1
Conjunctivitis (Eye disorders) | 1
Irritability (Psychiatric disorders) | 2
Belly twitch (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No